CLINICAL TRIAL: NCT00934531
Title: Can Cognitive Enhancers Reduce the Risk of Falls in Older People With Mild Cognitive Impairment? A Randomized Controled Trial
Brief Title: Donepezil and the Risk of Falls in Seniors With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Manuel Montero Odasso, Geriatrician/Clinician Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-09-427; 16086 (Other: REB)
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Falls; Gait; Balance; Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment (MCI); Falls; donepezil; gait variability
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil (Experimental): participants with MCI receiving donepezil
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator): Participants with MCI receiving placebo
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Participants with MCI will be randomized to either the experimental (donepezil) or placebo arm of the study.
  Experimental Arm: Participants with MCI will receive 5 mg/day of donepezil p.o. for 4 weeks, and thereafter 10 mg/day of donepezil p.o. for a period of 5 months, yielding a total period of intervention of 6 months from baseline.
  Placebo Arm: Participants with MCI will receive a matched placebo p.o. for 4 weeks, and thereafter will receive a new matched placebo p.o. for the next 5 months, yielding a total period of intervention of 6 months from baseline.
  Other Names: donepezil (Aricept)

SUMMARY:
Compared with cognitively normal older adults, those with mild cognitive problems (MCI) have a two-fold higher rate of falls, sustain more fractures, and have a higher rate of mortality due to falls. Why older adults with cognitive problems fall more frequently is not completely understood. What is known, however, is that attention is a necessary cognitive resource for normal walking and impairments in attention are associated with increased risk of falls in older adults.

It has been suggested that cholinesterase inhibitors (ChEI), medications used for treatment of dementia, may improve motor function and walking (gait performance). Since ChEI are known to improve attention, we hypothesized that ChEI will reduce falls risk in people with MCI by improving their gait velocity, improving their balance, and reducing their gait variability; a well-established risk factor for falls.

In the proposed study, we will evaluate the effect of donepezil (ChEI) on gait velocity, gait variability, and the balance on 140 elderly individuals with MCI (70 intervention and 70 controls). Gait variables will be measured using an electronic walkway, and balance confidence using a validated scale (Activities-Specific Balance Confidence Scale; ABC) over four months.

By characterizing and understanding the effects of cognitive enhancers on fall risk in older adults with cognitive impairments, we will be able to pave the way for a new approach to fall prevention in this population. We would establish that medications that augment cognitive function could be a complementary therapeutic option for reducing fall risk in people with MCI. This may lead to new approaches to prevent and treat fall risk in this population, which will lead to improve the autonomy and quality of life of seniors in early stage of dementia, and a decreased burden for the Ontario health care system.

DETAILED DESCRIPTION:
Older adults with cognitive problems have a higher risk of falls, with annual incidence of around 60-80%; at least twice that of cognitively normal older adults. The consequences of falls in this population can be quite serious; fallers with cognitive problems are approximately five times more likely to be admitted to institutional care than people with cognitive issues who do not fall. They are also at risk of major fall-related injuries such as fractures and head injuries leading to increased mortality. Although the reasons for the increased fall risk in cognitively impaired people are not completely understood, what is known is that these impaired cognitive abilities that can limit their attentional resource allocation while walking. As well, since executive function is also an important cognitive resource for normal walking performance, impairments in this domain are also associated with both dementia and risk of falls. Falls is a major cause of disability and dependence in older Ontarians, especially for those experiencing cognitive problems, and through their associated costs relating to hospital admissions, provision of treatments, and nursing home placements, forms a definite burden for the provincial health care system.

One approach that can be used to understand the risk of falls in people with memory problems is to target them in the early stages of cognitive decline. Mild Cognitive Impairment (MCI) is an entity that is conceived as a transitional state between benign age-related cognitive change and early dementia. Specific diagnostic criteria have been developed and validated to diagnose MCI, with the prevalence of the diagnosis being estimated at 19% among older adults, increasing to 29% in those over age 85. People with MCI have been found to have a 10 to 15 times higher risk of developing Alzheimer's disease (AD), as well as a higher risk of falling compared with age-matched controls.

Although walking has long been considered as primarily an automatic motor task, emerging evidence suggests that this view may be overly simplistic. Cognitive function may play a key role in the regulation of even routine walking, particularly in older adults. Attention is a necessary cognitive resource for maintaining normal walking and there is evidence that cognitive and attentional deficits are independently associated with postural instability, impairment in performing daily living activities, and future falls. The role of cognition in walking is even more marked in people with cognitive dysfunction, whose gait performance is affected by any extra cognitive load. A sensitive way to quantify gait performance is by assessing the gait variability. Gait variability is defined as the stride-to-stride variation in time, and quantifies the automaticity of gait, with greater variability indicating less rhythmicity and a more unstable gait pattern. Evaluating gait variability offers an accurate methodology to identify subtle changes on walking because of pathological conditions or disease. For instance, cognitively normal older adults have low gait variability; however, high gait variability has been described in Parkinson's disease, Alzheimer disease, and has been associated with high risk of future falls and mobility decline. Additionally, previous studies have demonstrated that gait variability may serve as a clinically relevant parameter in the evaluation of mobility, and may be a responsive measure for different interventions in fall prevention.

Cholinesterase inhibitors have been tried in MCI individuals with the goal to delay the progression to dementia. A recent RCT demonstrated that cognitive enhancers, specifically donepezil, might improve cognition in this population; however, the effect was weak and had questionable clinical significance. Currently, there is no indication to use cognitive enhancers to treat people with MCI with the goal of delaying or preventing further functional or mobility decline.

Recently, it has been suggested that ChEI may improve gait performance through an improvement in attentional resource allocation due to the fact that ChEI are known to improve attention and executive function. We will expect as a result of our intervention with donepezil during a 6 month period, a reduction of gait variability, an important marker of fall risk, through an improvement on cognition, namely attention an executive function

ELIGIBILITY:
Inclusion Criteria:

* Age 65-100
* Male or Female
* Having Mild Cognitive Impairment (diagnosed using criteria validated by Petersen et. al)
* Acceptable Body Mass Index (BMI) range: 18-30
* Acceptable blood pressure (Systolic: 110-160, Diastolic: 50-110)
* Able to walk independently 10 meters without any gait aid
* Able to travel to Aging Brain and Memory Clinic for the assessments

Exclusion Criteria:

* Unable to understand English
* Low body weight (less than 99lb/45kg)
* Possible diagnosis of Alzheimer's Disease
* Use of herbal preparations such as St. John's Wort and ginko biloba
* History of drug or alcohol abuse/dependence
* History of psychiatric illness within the last two years, including depression
* Parkinsonism or any neurological disorder with residual motor deficit (e.g.: stroke, epilepsy)
* Musculoskeletal disorder detected by clinical examination which affects gait performance
* Active osteoarthritis affecting the lower limbs (American College of Rheumatology criteria)
* Use of psychotropic medication, which can affect motor performance
* Use of an anticholinergic agent (benztropines), other acetylcholinesterase inhibitors or cholinergic agents (bethanechol)
* Depression (score above 8/15 on the Geriatric Depression Scale - GDS)
* Comorbidities which may contradict use of ChEIs
* History of chronic bradycardia or sick sinus syndrome
* Severe COPD and/or asthma
* History of seizure disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Improvements in gait performance (Combined outcome: increase in gait velocity-cm/second- and/or reduction in gait variability assessed as standard deviation (SD) and coefficient of variation (CoV). | 6 months

SECONDARY OUTCOMES:
Improvement in: 1. Balance confidence 2. Balance sway 3. Attention 4. Executive function 5. Reduction of number of Falls. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Montero Odasso, MD, PhD, Principal Investigator — The University of Western Ontario, Dept. of Medicine, Div. of Geriatric Medicine
Locations (1):
- St. Joseph's Health Care London, Parkwood Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Montero-Odasso M, Wells J, Borrie M. Can cognitive enhancers reduce the risk of falls in people with dementia? An open-label study with controls. J Am Geriatr Soc. 2009 Feb;57(2):359-60. doi: 10.1111/j.1532-5415.2009.02085.x. No abstract available. PMID 19207156
- [Background] Montero-Odasso M. The value of gait velocity test for high-function populations. J Am Geriatr Soc. 2006 Dec;54(12):1949-50; author reply 1950. doi: 10.1111/j.1532-5415.2006.00952.x. No abstract available. PMID 17198509
- [Background] Montero-Odasso M, Schapira M, Soriano ER, Varela M, Kaplan R, Camera LA, Mayorga LM. Gait velocity as a single predictor of adverse events in healthy seniors aged 75 years and older. J Gerontol A Biol Sci Med Sci. 2005 Oct;60(10):1304-9. doi: 10.1093/gerona/60.10.1304. PMID 16282564
- [Background] Montero-Odasso M, Speechley M, Chertkow H, Sarquis-Adamson Y, Wells J, Borrie M, Vanderhaeghe L, Zou GY, Fraser S, Bherer L, Muir-Hunter SW. Donepezil for gait and falls in mild cognitive impairment: a randomized controlled trial. Eur J Neurol. 2019 Apr;26(4):651-659. doi: 10.1111/ene.13872. Epub 2018 Dec 26. PMID 30565793
- [Derived] Montero-Odasso M, Wells JL, Borrie MJ, Speechley M. Can cognitive enhancers reduce the risk of falls in older people with mild cognitive impairment? A protocol for a randomised controlled double blind trial. BMC Neurol. 2009 Aug 12;9:42. doi: 10.1186/1471-2377-9-42. PMID 19674471